CLINICAL TRIAL: NCT01145768
Title: A Phase 1, Single Center, Double-blind, Randomized, Placebo- Controlled, Parallel-group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral TC-5214 (S-Mecamylamine) After Administration of Single and Multiple Ascending Doses for up to 8 Days in Healthy Male and Female Subjects
Brief Title: To Investigate the Safety and Tolerability of TC-5214 Following Oral Administration of Multiple Doses for up to 8 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4130C00006
Record Dates: First submitted 2010-06-07; First posted 2010-06-17 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Double-blind; randomized; placebo-controlled; parallel-group study; Safety; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Each cohort will have 9 volunteers that will receive TC-5214
  Interventions: Drug: TC-5214
- 2 (Placebo Comparator): Each cohort will have 3 volunteers that will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — 4 mg tablet, oral, BID, group 1
  Arms: 1
Drug: TC-5214 — TBD tablet, oral, BID, groups 2-6
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
To investigate the safety and tolerability of TC-5214 following oral administration of single and multiple ascending doses compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and nonpregnant, nonlactating female, with suitable veins for cannulation or repeated venipuncture
* Contraceptive use from the first dose of investigational product until12 weeks after their last dose
* Body mass index (BMI) between 19 and 32 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* History of any clinically significant medical, neurologic or psychiatric disease or disorder which, in the opinion of the Investigator and Sponsor, may either put the volunteer at risk because of participation in the study, or influence the results of
* History of gastrointestinal surgery (except for cholecystectomy and appendectomy) or unintentional rapid weight loss
* Volunteers with a history of suicide attempts in the past year and/or seen by the Investigator as having a significant history of risk of suicide or homicide, or considered at risk for suicide or homicide during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability assessed by incidence and severity of AE's, abnormalities in vital sign assessments, ECG's, telemetry, clinical lab assessments, physical exams, neurological exams, suicidality evaluations, visual acuity tests and digital ECGs | Collected prior to treatment, during treatment and for 7-10 days following discharge. Volunteers will be monitored througout the study for adverse events.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of TC-5214 in blood and urine after single and repeated oral doses by collecting blood and urine samples to measure drug concentration levels | Blood sampling, every in house day; urine collection ;Days -1 through Day 6, Days 8 through 11.
To assess the effect of food on the pharmacokinetics of TC-5214 following oral administration by collecting blood and urine samples to measure drug concentration levels. | Samples taken during the residential period at defined timepoints pre-dose and post-dose

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles, Inc.; Donna Holloway, Study Chair — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516